CLINICAL TRIAL: NCT01958411
Title: Correlation Between NAFLD, Epicardial Adipose Tissue and Vascular Inflammation Measured by Positron Emission Tomography (PET) With 18F-fluoro-deoxyglucose (FDG)
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: PET(NAFLD, EAT)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Atherosclerosis; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Atherosclerosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 18FDG-PET/CT

SUMMARY:
* Vascular inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis. 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques.
* Non-alcoholic fatty liver disease (NAFLD) is closely associated with many cardiometabolic risk factors. NAFLD can be detected by measuring liver fat accumulation using computed tomography (CT).
* Also epicardial adipose tissue (EAT) volume as determined by computed tomography (CT) is an independent marker of cardiovascular events in the general population.
* Therefore, the purpose of this investigators study is to compare the NAFLD severity and EAT volume with FDG uptake measured by PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Diabetes
* Stage 2 hypertension (resting blood pressure, ≥ 160/100 mmHg)
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect inflammation such as nonsteroidal antiinflammatory drug and statin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants who underwent a medical health check in the health promotion center in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Correlation between vascular inflammatory status measured by 18FDG PET and NAFLD measured by un-enhanced CT | 12 weeks
Correlation between vascular inflammatory status measured by 18FDG PET and epicardial adipose tissue measured by CT | 12 weeks

SECONDARY OUTCOMES:
The relationship of NAFLD with carotid intima media thickness | 12 weeks
The relationship of epicardial adipose tissue volume with carotid intima media thickness | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HJ, Lee CH, Kim S, Hwang SY, Hong HC, Choi HY, Chung HS, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Association between vascular inflammation and non-alcoholic fatty liver disease: Analysis by 18F-fluorodeoxyglucose positron emission tomography. Metabolism. 2017 Feb;67:72-79. doi: 10.1016/j.metabol.2016.11.004. Epub 2016 Nov 6. PMID 28081780